CLINICAL TRIAL: NCT01144065
Title: A Comparison of Hair Cortisol and Testosterone Levels in Patients With Acute MI and Controls With and Without Chronic Cardiovascular Disease or Diabetes
Brief Title: Hair Cortisol and Testosterone Levels in Patients With and Without Acute Myocardial Infarction(MI)
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HCT-1
Record Dates: First submitted 2010-06-07; First posted 2010-06-15 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial infarction; Cortisol; Testosterone
MeSH Terms: conditions — Myocardial Infarction | interventions — Testosterone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Heir samples for the measurement of cortisol and testosterone
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient with acute MI: Patients with acute MI ( elevated cardiac enzymes + chest pain or typical ECG changes)admitted to the cardiology department at Meir Medical Center
  Interventions: Procedure: Hair sampling for the measurement of cortisol and testosterone
- Patient with prior cardiovascular disease and/or diabetes: These patients do not have acute coronary syndrome or stroke. Prior cardiovascular disease (CVD) is defined as a history of hospital admission due to acute coronary artery occlusion, percutaneous coronary interventions (PCI), coronary artery bypass grafting, any aortic or peripheral vascular disease that was either symptomatic or required intervention, ischemic or hemorrhagic stroke or transient ischemic attack.
  Interventions: Procedure: Hair sampling for the measurement of cortisol and testosterone
- Patients without prior cardiovascular disease or diabetes: These patients do not have acute coronary syndrome or stroke Prior cardiovascular disease (CVD) or diabetes
  Interventions: Procedure: Hair sampling for the measurement of cortisol and testosterone

INTERVENTIONS:
Procedure: Hair sampling for the measurement of cortisol and testosterone — Hair sampling for the measurement of cortisol and testosterone

SUMMARY:
The purpose of this study is to determine whether hair levels of cortisol and testosterone are elevated in patients with acute MI compared to controls.

DETAILED DESCRIPTION:
Recently there has been a growing interest in measuring hair cortisol and testosterone levels. Hair grows approximately 1 centimeter per month, and hair analysis accurately reflects long-term endogenous production of these hormones. The association of elevated hair cortisol levels with chronic stress has been reported in several studies. Furthermore, we have recently demonstrated higher hair cortisol levels in patients admitted with acute myocardial infarction compared with patients admitted for other indications (the manuscript has recently been submitted for publication). Nevertheless it is still not clear whether hair cortisol levels are a risk factor for acute coronary event or for chronic cardiovascular diseases. In order to address this issue, further comparison of hair cortisol levels between patients with acute MI and a control group of patients with chronic cardiovascular diseases is needed.

Several studied have reported that endogenous testosterone concentrations are inversely associated with cardiovascular mortality and progression of atherosclerosis both in the coronary and the peripheral arteries. However these studies used a single serum testosterone level and therefore may not accurately represent the chronic endogenous production of this hormone. It may be that the association of testosterone levels and cardiovascular disease may be better evaluated using the hair technique. Nevertheless this association has not been studied yet.

Aim of the study:

To compare hair cortisol and testosterone levels in patients admitted with acute MI to stable patients with prior cardiovascular diseases or diabetes and patients with no history of cardiovascular diseases.

Secondary endpoint:

To evaluate the association between hair cortisol and testosterone with the burden of coronary atherosclerosis. The latter will be quantified only in the AMI patients undergoing coronary angiography by assessing the non culprit coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

General:

* Males
* Age>30

Cases:

* Patients with acute MI ( elevated cardiac enzymes + chest pain or typical ECG changes)

Control group 1:

Will include patients with at least 1 of the following:

* Prior cardiovascular disease (CVD). CVD is defined as a history of hospital admission due to acute coronary artery occlusion, percutaneous coronary interventions (PCI), coronary artery bypass grafting, any aortic or peripheral vascular disease that was either symptomatic or required intervention, ischemic or hemorrhagic stroke or transient ischemic attack.
* Diabetes mellitus. (Defined when it is reported by the patient or appears in his medical records, or if the patient has received regular treatment with oral hypoglycemic agents or insulin)

Control group 2:

* Patients without prior cardiovascular disease or diabetes mellitus (see definitions above).

Exclusion Criteria:

* Corticosteroid treatment in the last 12 months.
* Diagnosis of Cushing's or Addison's disease.
* Diagnosed hypogonadism treated with testosterone
* Dyed hair.
* Inability to sign inform consent.
* Any hospital admission during the 6 months prior to enrolment
* Morbid obesity (BMI>35)

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases:
  Patient with acute MI admitted to the cardiology department at Meir Medical Center
  Controls:
  Control group 1:
  patients with prior cardiovascular disease and/or diabetes:from intrnal medicine ward and the outpatient clinic
  Control group 2:
  Patients without prior cardiovascular disease or diabetes:from intrnal medicine ward and the outpatient clinic
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2010-08

PRIMARY OUTCOMES:
Comparison of hair cortisol and testosterone levels between the patients with acute MI and the 2 control groups | 1 day
  The study does not include a follow-up period

SECONDARY OUTCOMES:
Correlation of hair cortisol and testosterone with the burden of coronary atherosclerosis in the MI group | 1 day
  Coronary atherosclerosis will be quantitated in the MI patients that will undergo coronary angiography. We will evaluate the association of the atherosclerosis burden with Hair cortisol and testosterone levels

CONTACTS AND LOCATIONS:
Overall Officials: David Pereg, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

REFERENCES:
- [Background] Sauve B, Koren G, Walsh G, Tokmakejian S, Van Uum SH. Measurement of cortisol in human hair as a biomarker of systemic exposure. Clin Invest Med. 2007;30(5):E183-91. doi: 10.25011/cim.v30i5.2894. PMID 17892760
- [Background] Van Uum SH, Sauve B, Fraser LA, Morley-Forster P, Paul TL, Koren G. Elevated content of cortisol in hair of patients with severe chronic pain: a novel biomarker for stress. Stress. 2008 Nov;11(6):483-8. doi: 10.1080/10253890801887388. PMID 18609301
- [Background] Brotman DJ, Golden SH, Wittstein IS. The cardiovascular toll of stress. Lancet. 2007 Sep 22;370(9592):1089-100. doi: 10.1016/S0140-6736(07)61305-1. PMID 17822755
- [Background] Khaw KT, Dowsett M, Folkerd E, Bingham S, Wareham N, Luben R, Welch A, Day N. Endogenous testosterone and mortality due to all causes, cardiovascular disease, and cancer in men: European prospective investigation into cancer in Norfolk (EPIC-Norfolk) Prospective Population Study. Circulation. 2007 Dec 4;116(23):2694-701. doi: 10.1161/CIRCULATIONAHA.107.719005. Epub 2007 Nov 26. PMID 18040028
- [Background] Muller M, van den Beld AW, Bots ML, Grobbee DE, Lamberts SW, van der Schouw YT. Endogenous sex hormones and progression of carotid atherosclerosis in elderly men. Circulation. 2004 May 4;109(17):2074-9. doi: 10.1161/01.CIR.0000125854.51637.06. Epub 2004 Apr 19. PMID 15096452